CLINICAL TRIAL: NCT00667589
Title: Four-arm Study to Evaluate Urea 40% Cream, Fluocinonide 0.05% Cream, Tazarotene 0.1% Cream, and an Emollient Cream for the Treatment of Hand-foot Skin Reaction Related to the Use of Multi-targeted Tyrosine Kinase Inhibitor Sorafenib.
Brief Title: Sorafenib-induced Hand- Foot Skin Reaction Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted due to poor subject accrual.
Sponsor: Northwestern University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Dennis West, Professor in Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU2149
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Hand-foot Skin Reaction; Rash
Keywords: sorafenib; rash; hand foot skin reaction
MeSH Terms: conditions — Exanthema | interventions — Urea; Fluocinonide; tazarotene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- urea 40% cream (Experimental)
  Interventions: Drug: urea 40% cream
- fluocinonide 0.05% cream (Experimental)
  Interventions: Drug: fluocinonide 0.05% cream
- tazarotene 0.1% cream (Experimental)
  Interventions: Drug: tazarotene 0.1% cream
- bland emollient cream (Experimental)
  Interventions: Drug: bland emollient cream (Udderly smooth® Udder Cream)

INTERVENTIONS:
Drug: urea 40% cream — urea 40% cream applied twice per day to affected areas
  Other Names: carmol 40
  Arms: urea 40% cream
Drug: fluocinonide 0.05% cream — fluocinonide 0.05% cream applied twice per day to affected areas
  Arms: fluocinonide 0.05% cream
Drug: tazarotene 0.1% cream — tazarotene 0.1% cream applied twice per day to affected areas
  Other Names: tazarac
  Arms: tazarotene 0.1% cream
Drug: bland emollient cream (Udderly smooth® Udder Cream) — bland emollient cream applied twice per day to affected areas
  Other Names: Udderly smooth® Udder Cream
  Arms: bland emollient cream

SUMMARY:
The purpose of this study is to evaluate treatments for a rash caused by sorafenib.

DETAILED DESCRIPTION:
This study will compare compare the effectiveness of four creams (urea 40% cream, fluocinonide 0.05% cream, tazarotene 0.1% cream, and Udderly smooth® Udder Cream) in treating hand-foot skin reaction (HFSR), a rash caused by sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving sorafenib as monotherapy or in combination if other agents are not known to cause HFSR.
* Subjects must be 18 years or older.
* Patients must provide written informed consent to participate in the study.
* Women of childbearing potential and men must be willing to use an effective method of contraception while participating in this study and for at least two weeks after completing treatment in the study.
* Women in this study need to have a negative urine pregnancy test before starting study medications.

Exclusion Criteria:

* Patients simultaneously taking another anti-cancer agent or combination of anti-cancer agents known to cause hand foot syndrome (pegylated doxorubicin, 5-fluorouracil, cytarabine).
* Patients with an active dermatological condition due to previous chemotherapy or biologic therapy affecting the hands.
* Patients with pre-existing dermatological condition affecting the hands or feet.
* Women who have a positive pregnancy test or are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis West, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Udderly Smooth® Emollient: emollient applied twice per day to affected areas
Period: Overall Study
Arm/Group | Fluocinonide 0.05% Cream | Udderly Smooth® Emollient | Tazarotene 0.1% Cream | Urea 40% Cream
Started | 1 | 0 | 3 | 2
Completed | 0 | 0 | 0 | 1
Not Completed | 1 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluocinonide 0.05% Cream | Udderly Smooth® Emollient | Tazarotene 0.1% Cream | Urea 40% Cream | Total
Number analyzed (Participants) | 1 | 0 | 3 | 2 | 6
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0 | 0 | 0
  Between 18 and 65 years | 1 |  | 1 | 2 | 4
  >=65 years | 0 |  | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 61.0 (0) |  | 63.3 (12.7) | 60.5 (3.5) | 62.0 (9.3)
Gender [Number; unit: participants]
  Female | 0 |  | 2 | 2 | 4
  Male | 1 |  | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Skindex-16 Total Score Between Baseline and 8 Weeks
Description: The Skindex-16 questionnaire contains 16 questions related to quality of life in patients with skin disease. Total scores may range from 0 to 96, where 0 is associated with a better quality of life and 96 is associated with a worse quality of life. The data provided below indicates the change in the Skindex-16 total score between baseline and at 8 weeks.
Time Frame: baseline and 8 weeks
Population: Results for subjects from the fluocinonide 0.05% cream arm, subjects from the Tazarotene 0.1% cream arm, and one subject from the Urea 40% cream arm are not included in analysis because these subjects did not complete a Skindex-16 questionnaire at 8 weeks. No subjects were randomized to the Udderly Smooth Emollient arm.
Measure: Number; unit: units on a scale
Arm/Group | Urea 40% Cream
Number analyzed (Participants) | 1
units on a scale | -20

2. Secondary Outcome: Change in Skindex-16 Total Score Between Baseline and 2 Weeks
Description: The Skindex-16 questionnaire contains 16 questions related to quality of life in patients with skin disease. Total scores may range from 0 to 96, where 0 is associated with a better quality of life and 96 is associated with a worse quality of life. The data provided below indicates the change in the Skindex-16 total score between baseline and at 2 weeks.
Time Frame: baseline and 2 weeks
Population: Results for one subject from the Tazarotene 0.1% cream arm and one subject from the Urea 40% cream arm are not included in analysis because these subjects did not completed a Skindex-16 questionnaire at 2 weeks. No subjects were randomized to the Udderly Smooth Emollient arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluocinonide 0.05% Cream | Tazarotene 0.1% Cream | Urea 40% Cream
Number analyzed (Participants) | 1 | 2 | 1
units on a scale | 36 | -9.5 (12.0) | 1

ADVERSE EVENTS:
Arm/Group | Fluocinonide 0.05% Cream | Udderly Smooth® Emollient | Tazarotene 0.1% Cream | Urea 40% Cream
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes